CLINICAL TRIAL: NCT05808049
Title: A Randomized, Double Blind, Placebo Controlled Clinical Trial to Evaluate the Efficacy and Safety of MXP22 on Liver Health
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of MXP22 on Liver Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SY/211203/MASP/NFLD
Record Dates: First submitted 2023-02-14; First posted 2023-04-11 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Probiotics; Antioxidants; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sequentially numbered, sealed, opaque envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MXP22 (Probiotic and antioxidant capsule) (Experimental): Dose : NLT 4 Billion CFU/Capsule Route: Oral Administration Regimen: 1 capsule to be taken once daily after lunch for 120 days
  Interventions: Other: MXP22 (Probiotic and antioxidant capsule)
- Placebo (Microcrystalline Cellulose ) (Placebo Comparator): Dose : NLT 4 Billion CFU/Capsule Route: Oral Administration Regimen: 1 capsule to be taken once dailybafter lunch for 120 days
  Interventions: Other: Placebo (Microcrystalline Cellulose)

INTERVENTIONS:
Other: MXP22 (Probiotic and antioxidant capsule) — Dose: NLT 4 Billion CFU/Capsule Route: Oral Administration Regimen: 1 capsule to be taken once daily after lunch for 120 days
  Arms: MXP22 (Probiotic and antioxidant capsule)
Other: Placebo (Microcrystalline Cellulose) — Dose: NLT 4 Billion CFU/Capsule Route: Oral Administration Regimen: 1 capsule to be taken once daily after lunch for 120 days
  Arms: Placebo (Microcrystalline Cellulose )

SUMMARY:
A randomized, double blind, placebo controlled clinical trial to evaluate the efficacy and safety of MXP22 on liver health

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged more than equal to 30 and less than or equal to 60 years, diagnosed with NAFLD within last 2 years.
2. CAP scores more than equal to 248 and less than or equal to 270 dB/m indicating steatosis grade I/ II.
3. Non-alcoholics (little or no consumption of alcohol).
4. Willing to participate in the study with a signed and dated written consent.
5. Overweight and obese participant with BMI more than or equal to 25 kg/m2.
6. Having at least 3 of the following five metabolic risk factors:

i Waist circumference: Men: more than or equal to102 cm (40.15 inches); Women more than or equal to 88 cm (34.65 inches).

ii Triglycerides >150 mg/dL. iii Blood pressure more than or equal to 130 mm Hg (systolic, SBP) and/or more than or equal to 85 mm Hg (diastolic, DBP).

iv Fasting blood glucose more than or equal to 100 mg/ dl. v Low HDL level: Men: < 40 mg/dL; Women: < 50 mg/dL.

Exclusion Criteria:

1. Treatment of NAFLD for at least 3 months prior to the screening.
2. History of decompensated liver disease (ascites, encephalopathy, variceal bleeding).
3. Participants with liver cirrhosis, any concomitant liver disease.
4. Participants with systemic inflammatory disease or autoimmune disorders.
5. Participants with blood pressure Less than or equal to 160 mm Hg (systolic, SBP) and/or less than or equal to 95 mm Hg (diastolic, DBP).
6. Participants with Fasting blood glucose Less than or equal to 140 mg/ dl.
7. Participants with cardiopulmonary disease.
8. Heavy alcohol drinkers defined as follows:

   i For men, consuming more than 4 drinks on any day or more than 14 drinks/week ii For women, consuming more than 3 drinks on any day or more than 7 drinks/week
9. Participants with liver cancer - primary hepatocellular carcinoma or liver metastasis.
10. Participants with other systemic disorders of the heart, lungs, blood, and endocrine system, including thyroid dysfunction and Type I diabetes mellitus.
11. Histologic evidence of NASH with fibrosis stage (METAVIR score) F1 or F4.
12. Individuals with Inflammatory bowel diseases.
13. Use of medications containing systemic steroids, methotrexate corticosteroids, amiodarone, tamoxifen, valproate, vitamin E, omega-3, Anti-retroviral agents; 1 month prior to screening.
14. Intake of probiotics (lactic acid bacteria, etc.), prebiotics (dietary fiber, fructooligo saccharide, etc.), new biotics, fermented milk and proton pump inhibitor within one month before screening or during the study period.
15. Participants who have hypersensitivity to the test drug/ placebo or components contained in the test drug/placebo or have severe allergic reactions.
16. Females who are breast-feeding, lactating, pregnant or intending to become pregnant.
17. Regular use of a probiotic or prebiotic supplement within 3 months prior to screening.
18. Antibiotic use within 3 weeks prior to screening.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Fibroscan | Day 120.
  To evaluate the effect of 120 days consumption of MXP22 on hepatic steatosis as assessed by the change in Controlled Attenuation Parameter score on fibroscan from baseline to the end of the study, as compared to that in placebo

SECONDARY OUTCOMES:
AST & ALT | Day 0, 60 and 120
  Liver health as assessed by the significant change in the AST & ALT levels from baseline ascompared to that in placebo.
Lipid Profile | Day 0, 60 and 120
  Lipid profile as assessed by the significant change in the total Cholesterol, HDL Cholesterol, LDL Cholesterol and Triglycerides from baseline to end point in comparison to the placebo.
Inflammatory markers | Day 0 and 120
  The inflammatory factors as assessed by the change in Interlukins-6 and Tumour Necrosis Factor alpha from baseline to end point in comparison to the placebo.
serum Lipopolysaccharide level | Day 0 and 120
  On dietary endotoxemia as assessed by the significant change in the serum Lipopolysaccharide level after a high fat diet
Fibroscan | [Time Frame: Day 0, Day 60 and Day 120
  To evaluate the effect of 120 days consumption of MXP22 on hepatic steatosis as assessed by the change in Controlled Attenuation Parameter score on fibroscan from baseline to the end of the study, as compared to that in placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sudhir Maharshi, MBBS DNB Gastro, Principal Investigator — Dr. Sudhir Maharshi Gastro clinic
Locations (2):
- India (2):
  - JNU institute of medical science and research, Jaipur, Rajashthan
  - Dr. Sudhir Maharshi Gastro clinic, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided